CLINICAL TRIAL: NCT05716321
Title: Pain and Disability Outcomes in Post Amputation Patients
Status: Recruiting | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Sanjib D Adhikary, Professor of Anesthesiology,, Milton S. Hershey Medical Center
Other Study IDs: STUDY20483
Record Dates: First submitted 2023-01-05; First posted 2023-02-08 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Limb Pain, Phantom; Residual Limbs Pain; Disability Physical
Keywords: Amputation
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to evaluate efficacy of varied medical and procedural therapies used to treat pain after surgical amputation of a limb. The primary outcome will be assessment of pain severity at rest and with movement as measured by pain scores on Numerical Rating Scale (NRS) 0 to 10, where 0 is not pain and 10 is the worst pain possible, taken on post-operative day 1, day 7, 30 days, 90 days, 6 months, and 1 year (+/- 3 days at each time point).

DETAILED DESCRIPTION:
The objective of this study is to evaluate efficacy of varied medical and procedural therapies used to treat pain for surgical amputation of a limb.

At present there are number of different type of therapies are performed in the patients who is going through an amputation of any limb for management of their pain adequately such as peripheral nerve block, epidurals, peripheral nerve stimulators etc. However, the effects of these different procedures performed at different time intervals have not been evaluated for their effects on phantom pain and somatic pain long term after the procedures in these group of patients.

We will be collecting the following data from these patients to see if there is any particular intervention done at particular time of the procedure ( before the amputation vs. after the amputation) affect the long term outcome of these patients such as development of Phantom pain, or chronic pain

The primary outcome will be assessment of pain severity at rest and with movement as measured by pain scores on Numerical Rating Scale (NRS) 0 to 10, where 0 is not pain and 10 is the worst pain possible, taken on postoperative day 1, day 7, 30 days, 90 days, 6 months, and 1 year (+/- 3 days at each time point).

The secondary outcomes will be 1) phantom limb pain severity as rated on NRS 2) Residual limb (stump) pain as rated on NRS 3) phantom limb sensations 4) Pain Disability Index scores 5) Morphine milligram equivalents. These secondary outcomes will be assessed at the same intervals as the primary outcome.

This study will help us to find out if there is any utility of any of these procedures performed at particular time of the procedure helps them more than the others for development of somatic or phantom pain.

ELIGIBILITY:
Inclusion Criteria:

1. Ages between 18 and 89 years old, inclusive
2. Patients scheduled for surgical limb amputation at Penn State Hershey Medical Center

Exclusion Criteria:

1. Patients who cannot cooperate or consent
2. Patients who cannot understand or speak English
3. Patients with a history of chronic regional pain syndromes
4. Patients suffering from alcohol and/or drug abuse -based on previous Dx listed in the MRN
5. BMI >50

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for surgical limb amputation at Penn State Hershey Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Severity at rest and movement | 1 year
  The primary outcome will be assessment of pain severity at rest and with movement as measured by pain scores on Numerical Rating Scale (NRS) 0 to 10 taken on post-operative day 1, day 7, 30 days, 90 days, 6 months, and 1 year (+/- 3 days at each time point). 0 means no pain and 10 means the worst pain ever.

SECONDARY OUTCOMES:
Using NRS to rate phantom limb pain change in severity | 1 year
  The secondary outcomes will be phantom limb pain severity as rated on NRS. 0 to 10 taken on post-operative day 1, day 7, 30 days, 90 days, 6 months, and 1 year (+/- 3 days at each time point). 0 means no pain and 10 means the worst pain ever.
Using NRS to rate severity of change in pain | 1 year
  The third outcomes will be Residual limb (stump) pain as rated on NRS. 0 to 10 taken on post-operative day 1, day 7, 30 days, 90 days, 6 months, and 1 year (+/- 3 days at each time point). 0 means no pain and 10 means the worst pain ever.
Using NRS to rate of change in severity of Phantom limb sensations. | 1 year
  The fourth outcomes will be phantom limb sensations. 0 to 10 taken on post-operative day 1, day 7, 30 days, 90 days, 6 months, and 1 year (+/- 3 days at each time point). 0 means no sensation and 10 means the worst feeling ever.
Using NRS to rate Pain Disabiliy | 1 year
  The Fifth outcomes will be Pain Disability Index scores. 0 to 10 taken on post-operative day 1, day 7, 30 days, 90 days, 6 months, and 1 year (+/- 3 days at each time point). of 0 means no disability at all, and a score of 10 signifies that all of the activities in which you would normally be involved have been totally disrupted or prevented by your pain.
The amount of pain medication used. | 1 year
  The sixth outcomes will be the amount of Morphine milligram equivalents. The amount taken on post-operative day 1, Day 1 to day 7, day 8 to 30 days, 31 days to 90 days, 91 days to 6 months, and from 6 months to 1 year (+/- 3 days at each time point).

CONTACTS AND LOCATIONS:
Overall Officials: Sanjib Adhikary, M.B.B.S., MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
The IPD will be assigned a Study ID to protect the participants PHI. NO information will be shared with other investigators.